CLINICAL TRIAL: NCT04284410
Title: Integration of Prolonged Exposure (PE) and Coping Long-Term With Active Suicide Program (CLASP) for PTSD and Suicide Risk in Military Families
Brief Title: Integration of PE & Coping Long-Term With Active Suicide Program for PTSD & Suicide Risk in Military Families
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ronald E. Acierno, Visiting Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-1067
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Post Traumatic Stress Disorder; Suicidal Ideation
Keywords: depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLASP-PE arm (Experimental)
  Interventions: Behavioral: CLASP-PE arm

INTERVENTIONS:
Behavioral: CLASP-PE arm — Participants will complete 8-16 weekly or twice weekly individual therapy sessions (with total session number determined by clinical need, as is typical in clinical trials of PE for PTSD), 1 therapy session (session 3) with a supportive significant other (SO), consistent with the CLASP protocol, and 11 brief (30 minute) phone calls as possible, with calls occurring every week in between therapy sessions and on a less frequent basis following treatment termination up to 3 months after the final in-person therapy session. In addition, the supportive SOs will complete 11 brief (30 minute) phone calls with the therapist at the same frequency as participants. Participants will sign a release of information prior to involving the supportive significant other in treatment.

SUMMARY:
The purpose of this study is to develop an innovative, safe, acceptable, feasible, and efficacious integrated CLASP-PE intervention and to Collect pilot data to evaluate the preliminary evidence of the promise of the intervention. We hypothesize that the CLASP-PE intervention will demonstrate safety, acceptability, feasibility, and efficacy in the open trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in English. This is essential in order to complete the informed consent, self-report questionnaires, and homework assignments for the study.
* Diagnosis of PTSD according to the Clinician Administered PTSD Scale (CAPS). This is essential for the aims of the study, which include primarily to demonstrate a reduction in PTSD-related distress and ultimately in suicidal behaviors and thoughts.
* Suicidal ideation (SI) with a plan and/or a history of suicide attempts (SA). This is essential for the aims of the study, which include primarily to demonstrate a reduction in suicidal behaviors and thoughts as well as in PTSD related distress.
* Active duty service member
* Willingness to sign a release of information to allow for continuous communication between research study staff and treatment providers or between the research study staff and external mental health providers in order to ensure that any important information between the patient and their care team can be shared openly between the participating center and research staff involved in the patients care or assessment.

Exclusion Criteria:

* Current psychotic or manic episode as indicated by the MINI International Neuropsychiatric Interview. While it is possible that the intervention may be effective in individuals with psychosis, the research community needs to demonstrate the overall success of the intervention before it is applied to specialized subgroups, like individuals with psychosis. The intervention may also be eventually useful for individuals with a bipolar illness(defined by the presence of manic episodes) but likely that would require stabilization of mania prior to intervention implementation. As such these individuals will be excluded from the current study, though should possibly be included in future research depending on the results of the study.
* Current substance use disorder, severe (in the past terminology "dependence") that would preclude the ability to focus on PTSD and suicide symptom reduction. As with key exclusion criterion above, it is possible that individuals with a principal substance use disorder diagnosis may benefit from the intervention. However, the research community needs to demonstrate the overall success of the intervention (including in individuals with comorbid, but not principal) substance use disorders before it is applied in those with a principal substance use disorder.
* Current alternative evidence-based PTSD or suicide-focused individual psychotherapy, including current individual weekly Prolonged Exposure, current individual weekly Cognitive Processing Therapy, and current individual Coping LongTerm with Active Suicide Program (CLASP). Active involvement in an evidence-based PTSD or suicide-focused therapy would preclude the ability to scientifically test the effect of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a diagnosis of post-traumatic stress syndrome(PTSD)as assessed by The Clinician Administered PTSD Scale for DSM 5 (CAPS 5) | Baseline
  The CAPS 5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week.The CAPS-5 total score ranges from 0(absent) to 4(extreme/incapacitating)
Number of participants with a diagnosis of post-traumatic stress syndrome(PTSD)as assessed by The Clinician Administered PTSD Scale for DSM 5 (CAPS 5) | end of treatment (Upto 16 weeks from start of treatment)
  The CAPS 5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week.The CAPS-5 total score ranges from 0(absent) to 4(extreme/incapacitating)
Number of participants with a diagnosis of post-traumatic stress syndrome(PTSD)as assessed by The Clinician Administered PTSD Scale for DSM 5 (CAPS 5) | 3 months post treatment
  The CAPS 5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week.The CPAS-5 total score ranges from 0(absent) to 4(extreme/incapacitating)
Number of participants with a diagnosis of post-traumatic stress syndrome(PTSD)as assessed by The Clinician Administered PTSD Scale for DSM 5 (CAPS 5) | 6 months post treatment
  The CAPS 5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week.The CPAS-5 total score ranges from 0(absent) to 4(extreme/incapacitating)
The extent to which participants have been bothered by PTSD symptoms as assessed by the PTSD Checklist for DSM-5 (PCL-5) assessment. | Baseline
  The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The extent to which participants have been bothered by PTSD symptoms as assessed by the PTSD Checklist for DSM-5 (PCL-5) assessment. | before each session(participants will complete 8-16 weekly or twice weekly individual therapy sessions)
  The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The extent to which participants have been bothered by PTSD symptoms as assessed by the PTSD Checklist for DSM-5 (PCL-5) assessment. | end of treatment (Upto 16 weeks from start of treatment)
  The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The extent to which participants have been bothered by PTSD symptoms as assessed by the PTSD Checklist for DSM-5 (PCL-5) assessment. | 3 months post treatment
  The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The extent to which participants have been bothered by PTSD symptoms as assessed by the PTSD Checklist for DSM-5 (PCL-5) assessment. | 6 months post treatment
  The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
Number of patients with characteristic attitudes and symptoms of depression as measured by the Black depression Inventory (BDI) | Baseline
  The BDI is a 21-item self-report rating inventory that is rated in a 4 point scale from 0-3 based in severity with a maximum score if 63.
Number of patients with characteristic attitudes and symptoms of depression as measured by the Black depression Inventory (BDI) | before each session(participants will complete 8-16 weekly or twice weekly individual therapy sessions)
  The BDI is a 21-item self-report rating inventory that is rated in a 4 point scale from 0-3 based in severity with a maximum score if 63.
Number of patients with characteristic attitudes and symptoms of depression as measured by the Black depression Inventory (BDI) | end of treatment(Upto 16 weeks from start of treatment)
  The BDI is a 21-item self-report rating inventory that is rated in a 4 point scale from 0-3 based in severity with a maximum score if 63.
Number of patients with characteristic attitudes and symptoms of depression as measured by the Black depression Inventory (BDI) | 3 months post treatment
  The BDI is a 21-item self-report rating inventory that is rated in a 4 point scale from 0-3 based in severity with a maximum score if 63.
Number of patients with characteristic attitudes and symptoms of depression as measured by the Black depression Inventory (BDI) | 6 months post treatment
  The BDI is a 21-item self-report rating inventory that is rated in a 4 point scale from 0-3 based in severity with a maximum score if 63.
Severity of depression as assessed by the Quick Inventory of Depression Symptomatology (QIDS) The QIDS is a 16-item measure that is scored on a 4 point scale from 0-3 with a higher number indicating more severity of depression. | Baseline
Severity of depression as assessed by the Quick Inventory of Depression Symptomatology (QIDS) The QIDS is a 16-item measure that is scored on a 4 point scale from 0-3 with a higher number indicating more severity of depression. | before every session(participants will complete 8-16 weekly or twice weekly individual therapy sessions)
Severity of depression as assessed by the Quick Inventory of Depression Symptomatology (QIDS) The QIDS is a 16-item measure that is scored on a 4 point scale from 0-3 with a higher number indicating more severity of depression. | end of treatment (Upto 16 weeks from start of treatment)
Severity of depression as assessed by the Quick Inventory of Depression Symptomatology (QIDS) The QIDS is a 16-item measure that is scored on a 4 point scale from 0-3 with a higher number indicating more severity of depression. | 3 months post treatment
Severity of depression as assessed by the Quick Inventory of Depression Symptomatology (QIDS) The QIDS is a 16-item measure that is scored on a 4 point scale from 0-3 with a higher number indicating more severity of depression. | 6 months post treatment
Intensity of attitudes, behaviors and plans to commit suicide over the prior week as assessed by the Beck Scale for Suicidal ideation(BSSI) | Baseline
  BSSI is a 21-item self-report measure that is scored on a 3 point scale from 0-2 with a higher number indicting a greater suicidal ideation
Intensity of attitudes, behaviors and plans to commit suicide over the prior week as assessed by the Beck Scale for Suicidal ideation(BSSI) | end of treatment (Upto 16 weeks from start of treatment)
  BSSI is a 21-item self-report measure that is scored on a 3 point scale from 0-2 with a higher number indicting a greater suicidal ideation
Intensity of attitudes, behaviors and plans to commit suicide over the prior week as assessed by the Beck Scale for Suicidal ideation(BSSI) | 3 months post treatment
  BSSI is a 21-item self-report measure that is scored on a 3 point scale from 0-2 with a higher number indicting a greater suicidal ideation
Intensity of attitudes, behaviors and plans to commit suicide over the prior week as assessed by the Beck Scale for Suicidal ideation(BSSI) | 6 months post treatment
  BSSI is a 21-item self-report measure that is scored on a 3 point scale from 0-2 with a higher number indicting a greater suicidal ideation
Measure of suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline
  The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
Measure of suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | end of treatment (Upto 16 weeks from start of treatment)
  The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
Measure of suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | 3 months post-treatment
  The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
Measure of suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months post-treatment
  The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
Number of patients with anxiety, mood, psychotic, substance, and eating disorders as assessed by the MINI International Neuropsychiatric Interview (MINI) | Baseline
Extent to which client was satisfied with the training as assessed by the Client Satisfaction Questionnaire (CSQ) | end of treatment (Upto 16 weeks from start of treatment)
  The CSQ is an 8-item measure of client satisfaction rated on a 1-4 point Likert scale. A higher score indicates a higher satisfaction.
Feedback form participants as assessed by the Qualitative interview(QI) which will include a series of open ended questions aimed at eliciting feedback from participants about their perspective on the PE-CLASP Intervention | end of treatment (Upto 16 weeks from start of treatment)

SECONDARY OUTCOMES:
Number of potentially traumatic events in a respondent's lifetime as assessed by The Life Events Checklist for DSM-5 (LEC-5). | Baseline
  The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items. For each potentially traumatic life event, respondents rate their experience of that event on a 6-point nominal scale (1 = happened to me, 2 = witnessed it, 3 = learned about it, 4 = part of my job, 5 = not sure, and 6 = doesn't apply). The LEC-5 does not yield a total score or composite score.
Number of potentially traumatic events in a respondent's lifetime as assessed by The Life Events Checklist for DSM-5 (LEC-5). | end of treatment (Upto 16 weeks from start of treatment)
  The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items. For each potentially traumatic life event, respondents rate their experience of that event on a 6-point nominal scale (1 = happened to me, 2 = witnessed it, 3 = learned about it, 4 = part of my job, 5 = not sure, and 6 = doesn't apply). The LEC-5 does not yield a total score or composite score.
Number of potentially traumatic events in a respondent's lifetime as assessed by The Life Events Checklist for DSM-5 (LEC-5). | 3 months post treatment
  The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items. For each potentially traumatic life event, respondents rate their experience of that event on a 6-point nominal scale (1 = happened to me, 2 = witnessed it, 3 = learned about it, 4 = part of my job, 5 = not sure, and 6 = doesn't apply). The LEC-5 does not yield a total score or composite score.
Number of potentially traumatic events in a respondent's lifetime as assessed by The Life Events Checklist for DSM-5 (LEC-5). | 6 months post treatment
  The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items. For each potentially traumatic life event, respondents rate their experience of that event on a 6-point nominal scale (1 = happened to me, 2 = witnessed it, 3 = learned about it, 4 = part of my job, 5 = not sure, and 6 = doesn't apply). The LEC-5 does not yield a total score or composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Acierno, PhD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No